CLINICAL TRIAL: NCT03438630
Title: Health and Risk Factors in Patients With Hip and Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Linkoeping University (Other Government); Jonkoping County Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 160176
Record Dates: First submitted 2018-01-30; First posted 2018-02-20 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2021-10

CONDITIONS: Osteoarthritis
Keywords: socioeconomic factors; comorbidity; replacement surgery
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study cohort: All patients with a first registration (baseline) in the BOA Register between 2008 and 2016 (approximately n=75 000). These patients have sought treatment for knee and/or hip pain in primary health care in Sweden and been referred to the standardized core treatment of education and supervised exercises after confirmed clinical and/or radiographic OA diagnose.
- Control cohort: Covering the general Swedish population, who never have been included in the BOA register, will be recruited from the Swedish population register at Statistics Sweden and matched (1:3) to each patient in the study cohort by the same year of birth, gender and residence (as for the study cohort at baseline) (approximately n=225 000).

SUMMARY:
Hip and knee osteoarthritis is one of the leading causes of global disability. There is no cure for the disease, but research and guidelines recommends that patients with osteoarthritis, early after the diagnosis, receive individually adapted physical exercises, information about their disease and about self-management and, if needed, recommendations on weight loss as a core treatment to prevent disability and impairment in health. This core treatment improves symptoms in osteoarthritis by reducing pain and increasing function, and have the potential to delay replacement surgery. In Sweden, core treatment has since 2008, been standardized in a supported self-management programme and evaluation and follow-ups are registered in the National Quality Register BOA (Better management of patients with OsteoArthritis). The course of deterioration in pain and physical functioning among different individuals with osteoarthritis is currently difficult to predict. Factors such as socioeconomic status and comorbidity contribute to progression of the disease, but are not fully established. There is a need for early identification of individuals who have a good prognosis with slow disease development and those that should be recommended joint replacement surgery in the future. Overriding aim of the study is to increase knowledge about the population who has received education and supervised exercises as a core treatment for hip and knee osteoarthritis and been registered in the BOA Register and to identify factors that can predict long-term outcome for this population.

DETAILED DESCRIPTION:
Study design: This is a nationwide observational cohort study using prospectively obtained individual-level register data from five main sources; the BOA Register, the Swedish Hip Arthroplasty Register (SHAR), the Swedish Knee Arthroplasty Register (SKAR), Statistics Sweden and the National Board of Health and Welfare, Sweden. By using the personal identity number (PIN) that is unique to all citizens in Sweden, data will be merged together to create a research database that will be used for answering the following research questions in the study:

1. What are the differences between the population included in the BOA Register and the general Swedish population regarding health and socioeconomic factors?
2. What factors that predicts replacement surgery can be identified at the first registration, 3 months and/or 12 months follow-up, in the BOA Register in patients with hip or knee osteoarthritis?
3. What factors that predicts outcome after replacement surgery can be identified at the first registration, 3 months and/or 12 months follow-up in the BOA Register, in patients with hip or knee osteoarthritis?

Study population:The study cohort consists of all patients with a first registration (baseline) in the BOA Register between 2008 and 2016 (approximately n=75 000). These patients have sought treatment for knee and/or hip pain in primary health care in Sweden and been referred to the standardized core treatment of education and supervised exercises after confirmed clinical and/or radiographic osteoarthritis diagnose.

A control cohort (approximately n=225 000) covering the general Swedish population, who never have been included in the BOA register, will be recruited from the Swedish population register at Statistics Sweden and matched (1:3) to each patient in the study cohort by the same year of birth, gender and residence (as for the study cohort at baseline).

Data sources: In the study the investigators will collect the following data from the five registers: from the BOA Register: data reported by patients (e.g. most affected joint, pain, symptoms, health-related quality of life and physical activity level) and physiotherapists (e.g. earlier examinations and treatments) at baseline (the first registration before the standardized core treatment), and three and 12 months after. From the SHAR and the SKAR: patient-related and procedure-related data on all hip- and knee replacement surgeries in Sweden, including patient-reported outcomes (PROM) such as joint pain, health-related quality of life and satisfaction with treatment before surgery and one year postoperatively. From Statistics Sweden: data on socioeconomic factors and vital events such as birth, death, residence and marital status. From the National Board of Health and Welfare: data on comorbidity, health care consumption and expenditures of prescribed drugs.

ELIGIBILITY:
Inclusion Criteria: for participation in the standardized core treatment (of education and supervised exercises) and registration in the BOA Register are;

* pain from the knee or hip.
* diagnosis of osteoarthritis confirmed by a physical therapist, by medical history and a physical examination based on the clinical criteria for osteoarthritis

Exclusion Criteria: for participation in the standardized core treatment and registration in the BOA Register are;

* confirmed or suspicion of tumor, rheumatoid arthritis, sequel hip fracture, chronic pain or fibromyalgia,
* total joint replacement within the past 12 months,
* other surgery of the knee or hip joint within the past 3 months,
* not able to read or understand Swedish

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population who has received standardized core treatment of education and supervised exercises for hip and knee osteoarthritis and been registered in the BOA Register
Sampling Method: Non-Probability Sample
Enrollment: 288276 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Replacement surgery | up to the end of 2016
  Information from the SHAR and the SKAR Registers on eventual replacement surgery

SECONDARY OUTCOMES:
Socioeconomic factors - marital status | at baseline
  Data obtained from Statistics Sweden on marital status
Socioeconomic factors - education level | at baseline
  Data obtained from Statistics Sweden on education level
Socioeconomic factors - country of birth | at baseline
  Data obtained from Statistics Sweden on country of birth
Socioeconomic factors - occupation | at baseline
  Data obtained from Statistics Sweden on occupation
Socioeconomic factors - income | within three years prior to baseline
  Data obtained from Statistics Sweden on income
Socioeconomic factors - sick leave | within three years prior to baseline
  Data obtained from Statistics Sweden on sick leave
Consumption of drugs | within three years prior to baseline
  Data on expenditures of prescribed drugs from the Swedish Prescribed Drug Register at the National Board of Health Care, Sweden
Death | up to the end of 2016
  eventually registered as dead by Statistics Sweden
Comorbidity | within three years prior to baseline
  Data from the National Board of Health and Welfare on registered ICD10-codes
Health care consumption | within three years prior to baseline
  Data from the National Board of Health and Welfare on admission and discharge dates from health care units
Comorbidity | within three years prior to baseline
  Data from the National Board of Health and Welfare on registered classification of surgical interventions
Patient-reported outcome measure on most affected joint | at baseline, and at three and 12 months
  Data from the BOA Register on most affected joint
Patient-reported outcome measure on fear avoidance | at baseline, and at three and 12 months
  Data from the BOA Register on fear avoidance
Patient-reported outcome measure on physical activity | at baseline, and at three and 12 months
  Data from the BOA Register on physical activity level measured by questionnaire "In a typical week, how much time do you spend doing physical activity"
Patient-reported outcome measure on satisfaction with treatment | at baseline, and at three and 12 months
  Data from the BOA Register on satisfaction with treatment (the standardized core treatment) results measured by questionnaire
Patient-reported outcome measure musculoskeletal comorbidity | at baseline, and at three and 12 months
  Data from the BOA Register on musculoskeletal comorbidity measured in Charnley class (classifications of musculoskeletal impairment. Class A corresponds with unilateral hip or knee osteoarthritis (OA); Class B bilateral hip or knee OA; and Class C indicates multiple joint OA or some other condition that inhibits the patient's ability to walk)
Patient-reported outcome measure on pain | at baseline, and at three and 12 months
  Data from the BOA Register on pain in most affected joint, measured on VAS; (visual analogue scale) rating from 0-100, were 0 stands for no pain and 100 for maximum pain
Patient-reported outcome measure on health-related quality of life | at baseline, and at three and 12 months
  Data from the BOA Register on health-related quality of life measured by EuroQol 5-domain instrument (EQ-5D). The instrument consists of questions assessing 5 health outcome domains; mobility, self-care, usual activities, pain/discomfort and anxiety/ depression, and is summarized into a single score between 0 and 1 (full health). The instrument also includes a VAS assessing current overall health state scoring from 0 (worst imaginable health state) to 100 (best imaginable health state).
Patient-reported outcome measure on self-efficacy | at baseline, and at three and 12 months
  Data from the BOA Register on self-efficacy on ASES (Arthritis self-efficacy scale). ASES is a self-administered questionnaire which contains 11 items divided into 2 subgroups, self-efficacy pain and self-efficacy other symptoms. Each question is scored from 10 to 100, with "moderately certain" place midway between "very uncertain" and "very certain". Each subscale is scored separately, by taking the mean of the subscale items.
Physiotherapist-reported earlier examinations | at baseline and at three months
  Data from the BOA Register on earlier examinations of the affected joint prior to the standardized core treatment
Physiotherapist-reported earlier interventions | at baseline and at three months
  Data from the BOA Register on earlier interventions, prior to the standardized core treatment
Physiotherapist-reported compliance with intervention | at baseline and at three months
  Data from the BOA Register on compliance with the standardized core treatment intervention
Patient-reported outcome measures on satisfaction with treatment | before replacement surgery and at follow up one year
  Data from the SHAR and the SKAR Register on satisfaction with treatment (replacement surgery)
Patient-reported outcome measures - musculoskeletal comorbidity | before replacement surgery and at follow up one year
  Data from the SHAR and the SKAR Register on musculoskeletal comorbidity measured by Charnley class (Class A corresponds to unilateral hip/knee disease; Class B bilateral hip/knee disease; and Class C indicates multiple joint disease or some other condition that inhibits the patient's ability to walk).
Patient-reported outcome measures - pain | before replacement surgery and at follow up one year
  Data from the SHAR and the SKAR Register on pain from a VAS; visual analogue scale rating from 0-100, were 0 stands for no pain and 100 for maximum pain
Patient-reported outcome measures - health-related quality of life | before replacement surgery and at follow up one year
  Data from the SHAR and the SKAR Register on health-related quality of life measured by EuroQol 5-domain instrument (EQ-5D). The instrument consists of questions assessing 5 health outcome domains; mobility, self-care, usual activities, pain/discomfort and anxiety/ depression, and is summarized into a single score between 0 and 1 (full health). The instrument also includes a VAS assessing current overall health state scoring from 0 (worst imaginable health state) to 100 (best imaginable health state).

CONTACTS AND LOCATIONS:
Overall Officials: Ola Rolfson, Ass profess, Principal Investigator — Vastra Gotaland
Locations (1):
- Vastra Gotaland, Gothenburg, Sweden

REFERENCES:
- [Derived] Gustafsson K, Kvist J, Eriksson M, Rolfson O. What Factors Identified in Initial Osteoarthritis Management Are Associated With Poor Patient-reported Outcomes After THA? A Register-based Study. Clin Orthop Relat Res. 2023 Sep 1;481(9):1732-1742. doi: 10.1097/CORR.0000000000002681. Epub 2023 May 9. PMID 37159269
- [Derived] Gustafsson K, Kvist J, Eriksson M, Dell'Isola A, Zhou C, Dahlberg LE, Rolfson O. Health status of individuals referred to first-line intervention for hip and knee osteoarthritis compared with the general population: an observational register-based study. BMJ Open. 2021 Sep 13;11(9):e049476. doi: 10.1136/bmjopen-2021-049476. PMID 34518262
- [Derived] Gustafsson K, Rolfson O, Eriksson M, Dahlberg L, Kvist J. Study protocol for an observational register-based study on health and risk factors in patients with hip and knee osteoarthritis. BMJ Open. 2018 Oct 3;8(10):e022812. doi: 10.1136/bmjopen-2018-022812. PMID 30287673